CLINICAL TRIAL: NCT06474169
Title: Assessment of T-cell Response and In-vitro Proof-of-concept of T-cell Engineering in Chronic End-stage Kidney Disease Patients.
Brief Title: Assessment of T-cell Response and In-vitro Proof-of-concept of T-cell Engineering in Chronic ESKD Patients.
Acronym: LYMPHOVIRCT
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2023-11
Record Dates: First submitted 2024-06-10; First posted 2024-06-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Diseases
Keywords: end-stage kidney disease; T-cells response; Immunodeficiency; Proof of concept of T-cell therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For this study, the collection of blood samples is storage with specific samples :
  * Peripheral blood mononuclear cell (PBMC)
  * Serum
  * Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- n°1 (ESKD): end-stage chronic kidney disease
  Interventions: Other: 1 blood sample for each participant
- n°2 (stage 3 CKD): stage 3 chronic kidney disease
  Interventions: Other: 1 blood sample for each participant
- n°3 (healthy donors): healthy donors
  Interventions: Other: 1 blood sample for each participant

INTERVENTIONS:
Other: 1 blood sample for each participant — Blood sample for cohort n°1 and n°2 (collection during a peripheral venous blood sample, part of the standard of care for this disease) :
  1 blood sample for each patient 28mL of blood (4 tubes, 7mL per tube)
  Blood samples for cohort n°3 (collection during blood donation at Etablissement Français du Sang) :
  1 blood sample for each healthy donor 14mL of blood (2 tubes, 7mL per tube)

SUMMARY:
This is a comparative, prospective, non-interventional study to evaluate immune response in patients with chronic kidney disease. The primary objective is to define immunodeficiency (phenotype and function of T cells) in patients with end-stage kidney disease. The second objective is to provide an in-vitro proof-of-concept of T-cell engineering in the context of end-stage kidney disease.

The study population was patients with chronic kidney disease.

DETAILED DESCRIPTION:
The development of chronic kidney disease (CKD) and its progression to this terminal stage (end-stage kidney disease, ESKD) remains a significant source of reduced quality of life and premature mortality. ESKD represents the complete and definitive alteration of renal function requiring the use of renal replacement therapy (dialysis or kidney transplantation).

ESKD is associated with a significant increase in mortality, with a death rate of 10.9% and a median age of 77 years. Thus, the average survival of patients with ESKD is lower than that of the general population. Among the causes of death in ESKD, infectious diseases represent the 2nd cause of mortality and are responsible for 15 to 20% of deaths. The occurrence of complications increases with the decline of renal function, although individual risk remains poorly characterized. Thus, after infection, ESKD patients are at increased risk of complications, hospitalization, and death. This susceptibility to infections is explained by a complex alteration of the immune system, including a pro-inflammatory state and immunodeficiency. However, this immunodeficiency is still partially understood. Premature-aged T cells were found, with a decrease in naive T cells and an increase in memory T cells, suggesting a more advanced T-cell differentiation than in the population of the same age.

The study aims to describe immunodeficiency in patients with ESKD in order to better assess the infection risk for each patient, particularly in patients awaiting kidney transplantation.

This is a comparative, prospective, non-interventional study. Three groups of participants will be included: 1) patients with ESRK, 2) patients with stage 3 CKD, and 3) healthy donors. Participants will be included after being informed and after obtaining no opposition to participate. Immunodeficiency in patients with chronic kidney disease will be performed from a single blood sample.

A total of 100 participants will be included in this study based on the detection probability of naïve T cells (45% in patients with stage 3 CKD and healthy donors vs 10-15% in ESKD patients) and considered a power of 80% and an alpha risk of 5%.

The development of blood tests to evaluate the antiviral immune response could allow for the definition of new milestones for the development of future treatments or diagnostics for these diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Informed participants who did not object to participating in the study

Exclusion Criteria:

1. Chronic progressive infections
2. Prior organ transplantation (including bone marrow transplantation)
3. Previous treatment with immunosuppressive agents (such as Rituximab, Eculizumab, Tacrolimus or Ciclosporin, Cellcept or Imurel) within 2 years prior to inclusion
4. Participant under guardianship, curatorship or deprived of liberty
5. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease followed in Nephrology department of Orléans University Hospital (CHU d'Orléans):
  group 1 : end-stage kidney disease and group 2 : stage 3 chronic kidney disease
  Healthy donors in Etablissement français du Sang (EFS) in Orleans:
  Group 3 : healthy donors
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is to characterize T cell immunodeficiency in our cohort of end-stage kidney disease patients from a phenotypic and functional point of view. | Duration of blood collection (approximately 5 minutes in inclusion)
  Identify T cells and perform extensive phenotype. This analysis will be performed on mononuclear cells with a clinical flow cytometry system (panel of specific fluorophores will be used).
The primary outcome is to characterize T cell immunodeficiency in our cohort of end-stage kidney disease patients from a phenotypic and functional point of view. | Duration of blood collection (approximately 5 minutes in inclusion)
  Perform a non-specific assessment of T-cell activation in measuring the production of ATP ( adenosine triphosphate) and cytokines.
The primary outcome is to characterize T cell immunodeficiency in our cohort of end-stage kidney disease patients from a phenotypic and functional point of view. | Duration of blood collection (approximately 5 minutes in inclusion)
  Functional evaluation of T cells with specific viral assessment. Differents tests will be performed after peptidic stimulations: quantification of cytokines and proliferative capacities.

SECONDARY OUTCOMES:
in-vitro proof-of-concept of T-cell engineering | For each outcome, duration of blood collection (approximately 5 minutes in inclusion)
  Development of mRNA delivery system to restore T-cell function in ESKD patients through T-cell therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Center Hospitalier Universitaire d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishigami J, Matsushita K. Clinical epidemiology of infectious disease among patients with chronic kidney disease. Clin Exp Nephrol. 2019 Apr;23(4):437-447. doi: 10.1007/s10157-018-1641-8. Epub 2018 Sep 3. PMID 30178234
- [Background] Syed-Ahmed M, Narayanan M. Immune Dysfunction and Risk of Infection in Chronic Kidney Disease. Adv Chronic Kidney Dis. 2019 Jan;26(1):8-15. doi: 10.1053/j.ackd.2019.01.004. PMID 30876622
- [Background] Betjes MG. Immune cell dysfunction and inflammation in end-stage renal disease. Nat Rev Nephrol. 2013 May;9(5):255-65. doi: 10.1038/nrneph.2013.44. Epub 2013 Mar 19. PMID 23507826
- [Background] Betjes MG, Huisman M, Weimar W, Litjens NH. Expansion of cytolytic CD4+CD28- T cells in end-stage renal disease. Kidney Int. 2008 Sep;74(6):760-7. doi: 10.1038/ki.2008.301. Epub 2008 Jul 9. PMID 18615000
- [Background] Betjes MG, Langerak AW, van der Spek A, de Wit EA, Litjens NH. Premature aging of circulating T cells in patients with end-stage renal disease. Kidney Int. 2011 Jul;80(2):208-17. doi: 10.1038/ki.2011.110. Epub 2011 Apr 27. PMID 21525849
- [Background] Litjens NH, van Druningen CJ, Betjes MG. Progressive loss of renal function is associated with activation and depletion of naive T lymphocytes. Clin Immunol. 2006 Jan;118(1):83-91. doi: 10.1016/j.clim.2005.09.007. Epub 2005 Oct 27. PMID 16257266
- [Background] Xiang F, Chen R, Cao X, Shen B, Chen X, Ding X, Zou J. Premature aging of circulating T cells predicts all-cause mortality in hemodialysis patients. BMC Nephrol. 2020 Jul 13;21(1):271. doi: 10.1186/s12882-020-01920-8. PMID 32660510